CLINICAL TRIAL: NCT02274636
Title: Study of a Dietary Supplement for Reflux During Sleep
Acronym: SXDSFRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oral Care Research Associates, Seattle (Other)
Responsible Party: Principal Investigator, Jeff Burgess DDS MSD, Research Coordinator, Oral Care Research Associates, Seattle
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1401
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Xylitol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Data collection (No Intervention): This first phase will involve having you report to the research coordinator through email the presence or absence of several symptoms associated with GERD that can occur during sleep. Phase 1 will occur over 14 days (and nights).
- Intervention (Active Comparator): In the second phase of the study, each subject will be given either a gel containing xylitol or discs containing xylitol to use for 14 days (the duration of the second phase of the study). If given the gel, a small amount (specified in the directions) is to be applied to the mouth lining just before bed. If given the discs, one will be placed on the gums beside a molar in each cheek each night just before bed (specified in the directions). Each subject will be asked to continue to provide daily email communication with the research coordinator detailing symptoms suggesting reflux experienced the prior night during product use as was provided during phase 1 of the study.
  Interventions: Dietary Supplement: Xylitol

INTERVENTIONS:
Dietary Supplement: Xylitol — A comparison between discs and gel
  Arms: Intervention

SUMMARY:
This research study is a randomized, controlled study developed to test how well a dry mouth product that contains xylitol affects some of the symptoms of gastroesophageal reflux disease (GERD. Individuals who experience symptoms of gastro esophageal reflux disease (GERD) and who are accepted into the study will be asked to report on the frequency and severity of several symptoms specific to the condition that occur during sleep. The study is composed of two phases:

Phase one involves collection of baseline information for two weeks. Phase two is the intervention phase of the study. In this phase of the study, each subject will be randomly assigned (like flipping a coin) to use either "the product" of interest or a different dry mouth product for two weeks.

DETAILED DESCRIPTION:
The study is composed of two phases:

Phase one involves collection of baseline information for two weeks. Phase two is the intervention phase of the study. In this phase of the study, each subject will be randomly assigned (like flipping a coin) to use either "the product" of interest or a different dry mouth product for two weeks.

Phase 1

This first phase will involve having you report to the research coordinator through email the presence or absence of several symptoms associated with GERD that can occur during sleep. Phase 1 will occur over 14 days (and nights). You will also be asked to rate the relative severity of some of the symptoms. The information collected during this initial phase of the study will then be used to establish baseline values for the symptoms of interest and determine your eligibility for the intervention phase (phase 2) of the study.

Phase 2

In the second phase of the study, you will be given either enough gel or enough discs to use for 14 days (the duration of the second phase of the study). If you are given the gel, a small amount (specified in the directions) is to be applied to the mouth lining just before bed. If you are given the discs, one will be placed on the gums beside a molar in each cheek each night just before bed (specified in the directions). You will be asked to continue to provide daily email communication with the research coordinator detailing symptoms suggesting reflux experienced the prior night during product use as you did during phase 1 of the study.

During phases 1 and 2 of the study, you will be asked to continue taking any previously prescribed medication or over-the-counter preparations that you normally take for reflux and to maintain your regular dietary habits. However, you should not take any dry mouth remedy other than those supplied by the research coordinator just before bed.

ELIGIBILITY:
Inclusion Criteria:

1. A medical diagnosis of GERD
2. Awakening with a taste of refluxed stomach acid in the mouth
3. Heartburn during sleep
4. Voice hoarseness upon awakening
5. Antacid use at night
6. Dry mouth at bedtime or during the night
7. Experience difficulty chewing, swallowing, and speaking because of dry mouth

Exclusion Criteria:

1. Under 18
2. Prior history of any of these conditions:

   1. coronary artery disease
   2. gallbladder disease
   3. gastric or esophageal cancer
   4. peptic ulcer disease
   5. esophagitis, whether eosinophilic, infectious, or pill based
   6. esophageal motility disorders
3. A history of thoracic, esophageal, or gastric surgery
4. No medical examination in the prior year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Reduction in symptoms associated with GERD | two weeks
  Email questionnaire containing 9 questions of interest

CONTACTS AND LOCATIONS:
Overall Officials: Jeff A Burgess, DDS MSD, Study Director — Oral Care Research Associates, Seattle

REFERENCES:
- [Background] Holtmann G. Reflux disease: the disorder of the third millennium. Eur J Gastroenterol Hepatol. 2001 May;13 Suppl 1:S5-11. PMID 11430509
- [Background] Jung HK, Choung RS, Talley NJ. Gastroesophageal reflux disease and sleep disorders: evidence for a causal link and therapeutic implications. J Neurogastroenterol Motil. 2010 Jan;16(1):22-9. doi: 10.5056/jnm.2010.16.1.22. Epub 2010 Jan 31. PMID 20535322
- [Background] Ranjitkar S, Smales RJ, Kaidonis JA. Oral manifestations of gastroesophageal reflux disease. J Gastroenterol Hepatol. 2012 Jan;27(1):21-7. doi: 10.1111/j.1440-1746.2011.06945.x. PMID 22004279
- [Background] Bardhan KD, Strugala V, Dettmar PW. Reflux revisited: advancing the role of pepsin. Int J Otolaryngol. 2012;2012:646901. doi: 10.1155/2012/646901. Epub 2011 Nov 10. PMID 22242022
- [Background] Fass R, Pulliam G, Johnson C, Garewal HS, Sampliner RE. Symptom severity and oesophageal chemosensitivity to acid in older and young patients with gastro-oesophageal reflux. Age Ageing. 2000 Mar;29(2):125-30. doi: 10.1093/ageing/29.2.125. PMID 10791446
- [Background] Chait MM. Gastroesophageal reflux disease: Important considerations for the older patients. World J Gastrointest Endosc. 2010 Dec 16;2(12):388-96. doi: 10.4253/wjge.v2.i12.388. PMID 21191512
- [Background] Saritas Yuksel E, Vaezi MF. New developments in extraesophageal reflux disease. Gastroenterol Hepatol (N Y). 2012 Sep;8(9):590-9. PMID 23483833
- [Background] DeVault KR, Castell DO; American College of Gastroenterology. Updated guidelines for the diagnosis and treatment of gastroesophageal reflux disease. Am J Gastroenterol. 2005 Jan;100(1):190-200. doi: 10.1111/j.1572-0241.2005.41217.x. PMID 15654800
- [Background] Kahrilas PJ, Shaheen NJ, Vaezi MF, Hiltz SW, Black E, Modlin IM, Johnson SP, Allen J, Brill JV; American Gastroenterological Association. American Gastroenterological Association Medical Position Statement on the management of gastroesophageal reflux disease. Gastroenterology. 2008 Oct;135(4):1383-1391, 1391.e1-5. doi: 10.1053/j.gastro.2008.08.045. No abstract available. PMID 18789939
- [Background] Dolder M, Tutuian R. Laboratory based investigations for diagnosing gastroesophageal reflux disease. Best Pract Res Clin Gastroenterol. 2010 Dec;24(6):787-98. doi: 10.1016/j.bpg.2010.10.005. PMID 21126694
- [Background] Katz PO, Gerson LB, Vela MF. Guidelines for the diagnosis and management of gastroesophageal reflux disease. Am J Gastroenterol. 2013 Mar;108(3):308-28; quiz 329. doi: 10.1038/ajg.2012.444. Epub 2013 Feb 19. No abstract available. PMID 23419381
- [Background] Locke GR 3rd, Talley NJ, Fett SL, Zinsmeister AR, Melton LJ 3rd. Prevalence and clinical spectrum of gastroesophageal reflux: a population-based study in Olmsted County, Minnesota. Gastroenterology. 1997 May;112(5):1448-56. doi: 10.1016/s0016-5085(97)70025-8. PMID 9136821
- [Background] Fass R, Achem SR, Harding S, Mittal RK, Quigley E. Review article: supra-oesophageal manifestations of gastro-oesophageal reflux disease and the role of night-time gastro-oesophageal reflux. Aliment Pharmacol Ther. 2004 Dec;20 Suppl 9:26-38. doi: 10.1111/j.1365-2036.2004.02253.x. PMID 15527462
- [Background] Eckley CA, Rios Lda S, Rizzo LV. Salivary egf concentration in adults with reflux chronic laryngitis before and after treatment: preliminary results. Braz J Otorhinolaryngol. 2007 Mar-Apr;73(2):156-60. doi: 10.1016/s1808-8694(15)31060-0. PMID 17589721
- [Background] Guare RO, Ferreira MC, Leite MF, Rodrigues JA, Lussi A, Santos MT. Dental erosion and salivary flow rate in cerebral palsy individuals with gastroesophageal reflux. J Oral Pathol Med. 2012 May;41(5):367-71. doi: 10.1111/j.1600-0714.2011.01112.x. Epub 2011 Nov 14. PMID 22077728
- [Background] Wong WM, Lam KF, Cheng C, Hui WM, Xia HH, Lai KC, Hu WH, Huang JQ, Lam CL, Chan CK, Chan AO, Lam SK, Wong BC. Population based study of noncardiac chest pain in southern Chinese: prevalence, psychosocial factors and health care utilization. World J Gastroenterol. 2004 Mar 1;10(5):707-12. doi: 10.3748/wjg.v10.i5.707. PMID 14991943
- [Background] Jansson C, Nordenstedt H, Wallander MA, Johansson S, Johnsen R, Hveem K, Lagergren J. A population-based study showing an association between gastroesophageal reflux disease and sleep problems. Clin Gastroenterol Hepatol. 2009 Sep;7(9):960-5. doi: 10.1016/j.cgh.2009.03.007. Epub 2009 Mar 13. PMID 19286481
- [Background] Gisbert JP, Cooper A, Karagiannis D, Hatlebakk J, Agreus L, Jablonowski H, Zapardiel J. Impact of gastroesophageal reflux disease on patients' daily lives: a European observational study in the primary care setting. Health Qual Life Outcomes. 2009 Jul 2;7:60. doi: 10.1186/1477-7525-7-60. PMID 19573227
- [Background] Ferrus JA, Zapardiel J, Sobreviela E; SYMPATHY I study group. Management of gastroesophageal reflux disease in primary care settings in Spain: SYMPATHY I study. Eur J Gastroenterol Hepatol. 2009 Nov;21(11):1269-78. doi: 10.1097/MEG.0b013e32832a7d9b. PMID 19474743
- [Background] Gerson LB, Fass R. A systematic review of the definitions, prevalence, and response to treatment of nocturnal gastroesophageal reflux disease. Clin Gastroenterol Hepatol. 2009 Apr;7(4):372-8; quiz 367. doi: 10.1016/j.cgh.2008.11.021. Epub 2008 Dec 3. PMID 19111949
- [Background] Hungin AP, Hill C, Raghunath A. Systematic review: frequency and reasons for consultation for gastro-oesophageal reflux disease and dyspepsia. Aliment Pharmacol Ther. 2009 Aug 15;30(4):331-42. doi: 10.1111/j.1365-2036.2009.04047.x. PMID 19660016
- [Background] Wallander MA, Johansson S, Ruigomez A, Garcia Rodriguez LA, Jones R. Dyspepsia in general practice: incidence, risk factors, comorbidity and mortality. Fam Pract. 2007 Oct;24(5):403-11. doi: 10.1093/fampra/cmm050. Epub 2007 Aug 28. PMID 17728288
- [Background] Kusano M, Kouzu T, Kawano T, Ohara S. Nationwide epidemiological study on gastroesophageal reflux disease and sleep disorders in the Japanese population. J Gastroenterol. 2008;43(11):833-41. doi: 10.1007/s00535-008-2235-0. Epub 2008 Nov 18. PMID 19012036
- [Background] Fass R, Quan SF, O'Connor GT, Ervin A, Iber C. Predictors of heartburn during sleep in a large prospective cohort study. Chest. 2005 May;127(5):1658-66. doi: 10.1378/chest.127.5.1658. PMID 15888843
- [Background] Mody R, Bolge SC, Kannan H, Fass R. Effects of gastroesophageal reflux disease on sleep and outcomes. Clin Gastroenterol Hepatol. 2009 Sep;7(9):953-9. doi: 10.1016/j.cgh.2009.04.005. Epub 2009 Apr 16. PMID 19375520
- [Background] Marsicano JA, de Moura-Grec PG, Bonato RC, Sales-Peres Mde C, Sales-Peres A, Sales-Peres SH. Gastroesophageal reflux, dental erosion, and halitosis in epidemiological surveys: a systematic review. Eur J Gastroenterol Hepatol. 2013 Feb;25(2):135-41. doi: 10.1097/MEG.0b013e32835ae8f7. PMID 23111415
- [Background] Yoshikawa H, Furuta K, Ueno M, Egawa M, Yoshino A, Kondo S, Nariai Y, Ishibashi H, Kinoshita Y, Sekine J. Oral symptoms including dental erosion in gastroesophageal reflux disease are associated with decreased salivary flow volume and swallowing function. J Gastroenterol. 2012 Apr;47(4):412-20. doi: 10.1007/s00535-011-0515-6. Epub 2011 Dec 27. PMID 22200941
- [Background] Correa MC, Lerco MM, Cunha Mde L, Henry MA. Salivary parameters and teeth erosions in patients with gastroesophageal reflux disease. Arq Gastroenterol. 2012 Jul-Sep;49(3):214-8. doi: 10.1590/s0004-28032012000300009. PMID 23011245
- [Background] Fass R, Ofman JJ, Sampliner RE, Camargo L, Wendel C, Fennerty MB. The omeprazole test is as sensitive as 24-h oesophageal pH monitoring in diagnosing gastro-oesophageal reflux disease in symptomatic patients with erosive oesophagitis. Aliment Pharmacol Ther. 2000 Apr;14(4):389-96. doi: 10.1046/j.1365-2036.2000.00733.x. PMID 10759617
- [Background] Kao CH, Ho YJ, ChangLai SP, Liao KK. Evidence for decreased salivary function in patients with reflux esophagitis. Digestion. 1999;60(3):191-5. doi: 10.1159/000007658. PMID 10343131
- [Background] Helm JF, Dodds WJ, Hogan WJ. Salivary response to esophageal acid in normal subjects and patients with reflux esophagitis. Gastroenterology. 1987 Dec;93(6):1393-7. doi: 10.1016/0016-5085(87)90270-8. PMID 3678754
- [Background] Pope CE 2nd. Acid-reflux disorders. N Engl J Med. 1994 Sep 8;331(10):656-60. doi: 10.1056/NEJM199409083311007. No abstract available. PMID 8052276
- [Background] Smith DJ, Joshipura K, Kent R, Taubman MA. Effect of age on immunoglobulin content and volume of human labial gland saliva. J Dent Res. 1992 Dec;71(12):1891-4. doi: 10.1177/00220345920710120701. PMID 1452889
- [Background] Iorgulescu G. Saliva between normal and pathological. Important factors in determining systemic and oral health. J Med Life. 2009 Jul-Sep;2(3):303-7. PMID 20112475
- [Background] Helm JF, Dodds WJ, Hogan WJ, Soergel KH, Egide MS, Wood CM. Acid neutralizing capacity of human saliva. Gastroenterology. 1982 Jul;83(1 Pt 1):69-74. No abstract available. PMID 7075945
- [Background] http://www.moderndentistrymedia.com/jan_feb2012/walsh.pdf; Author: LJ Walsh; Title: Clinical aspects of salivary biology for the dental clinician. In ModerDentistryMedia
- [Background] Dutta SK, Agrawal K, Mahmoud MA. Modulation of salivation and heartburn in response to the site of acid infusion in the human oesophagus. Aliment Pharmacol Ther. 2010 Sep;32(6):795-800. doi: 10.1111/j.1365-2036.2010.04397.x. PMID 20629975
- [Background] Haag S, Holtmann G. Onset of relief of symptoms of gastroesophageal reflux disease: post hoc analysis of two previously published studies comparing pantoprazole 20 mg once daily with nizatidine or ranitidine 150 mg twice daily. Clin Ther. 2010 Apr;32(4):678-90. doi: 10.1016/j.clinthera.2010.03.020. PMID 20435237
- [Background] Armstrong D, Pare P, Pericak D, Pyzyk M; Canadian Pantoprazole GERD Study Group. Symptom relief in gastroesophageal reflux disease: a randomized, controlled comparison of pantoprazole and nizatidine in a mixed patient population with erosive esophagitis or endoscopy-negative reflux disease. Am J Gastroenterol. 2001 Oct;96(10):2849-57. doi: 10.1111/j.1572-0241.2001.4237_a.x. PMID 11695354
- [Background] Vela MF. Medical treatments of GERD: the old and new. Gastroenterol Clin North Am. 2014 Mar;43(1):121-33. doi: 10.1016/j.gtc.2013.12.001. Epub 2013 Dec 31. PMID 24503363
- [Background] Burgess J, Lee P. XyliMelts time-release adhering discs for night-time oral dryness. Int J Dent Hyg. 2012 May;10(2):118-21. doi: 10.1111/j.1601-5037.2011.00532.x. Epub 2011 Oct 31. PMID 22040224
- [Background] Kerr AR, Corby PM, Shah SS, Epler M, Fisch GS, Norman RG. Use of a mucoadhesive disk for relief of dry mouth: a randomized, double-masked, controlled crossover study. J Am Dent Assoc. 2010 Oct;141(10):1250-6. doi: 10.14219/jada.archive.2010.0053. PMID 20884928
- [Background] Nwokediuko SC. Current trends in the management of gastroesophageal reflux disease: a review. ISRN Gastroenterol. 2012;2012:391631. doi: 10.5402/2012/391631. Epub 2012 Jul 11. PMID 22844607
- [Background] Helm JF, Dodds WJ, Pelc LR, Palmer DW, Hogan WJ, Teeter BC. Effect of esophageal emptying and saliva on clearance of acid from the esophagus. N Engl J Med. 1984 Feb 2;310(5):284-8. doi: 10.1056/NEJM198402023100503. PMID 6690951
- [Background] Printza A, Speletas M, Triaridis S, Wilson J. Is pepsin detected in the saliva of patients who experience pharyngeal reflux? Hippokratia. 2007 Jul;11(3):145-9. PMID 19582210